CLINICAL TRIAL: NCT05874219
Title: The Effect of Mupirocin 2% Ointment on the Duration of Stay of Temporary Hemodialysis Catheter Compared to Other Spray Antibiotics
Brief Title: Mupirocin 2% Ointment Vs Spray Antibiotics on Temporary Hemodialysis Catheter
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Salah ElDin Diab ELBohy, Assistant professor, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU R85/2023
Record Dates: First submitted 2023-04-25; First posted 2023-05-24 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Hemodialysis Complication; Hemodialysis Catheter Infection
MeSH Terms: interventions — Bacitracin; Mupirocin; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local antibiotic spray (Experimental): Local antibiotic spray (n=75) The intervention Sprayed 1 to 3 times /day for 45 day Neomycin sulphate 165,000 IU + Bacitracin zinc 12,500 IU Bivatracin Spray
  Interventions: Drug: Local antibiotic spray Neomycin sulphate 165,000 IU + Bacitracin zinc 12,500 IU
- Mupirocin 2% ointment (Active Comparator): (The standard) 10 mm of mupirocin ointment squeezed directly on to their exit sites from a 15 g tube with an outlet diameter of 5 mm mupirocin 2% ointment
  Interventions: Drug: Mupirocin 2% ointment

INTERVENTIONS:
Drug: Local antibiotic spray Neomycin sulphate 165,000 IU + Bacitracin zinc 12,500 IU — The intervention Sprayed 1 to 3 times /day
  Other Names: BIVATRACIN
  Arms: Local antibiotic spray
Drug: Mupirocin 2% ointment — 10 mm of mupirocin ointment squeezed directly on to their exit sites from a 15 g tube with an outlet diameter of 5 mm
  Arms: Mupirocin 2% ointment

SUMMARY:
In dialysis centers, many patients are undergoing hemodialysis simultaneously, which facilitates the spread of microorganisms by direct or indirect contact through the devices, equipment, surface contact, and hands of health profession Over time, catheters are prone to higher rates of infection, thrombosis, and central venous stenosis, it has also been shown that catheters are an independent (of infection) inflammatory stressor and lead to increased morbidity .

Catheters are aptly referred to as a bacterial highway, and a biofilm formation around the catheter is often the breeding ground of bacteria and fungi, which can easily spread to the bloodstream Infectious complications are the most serious with regards to patient morbidity and mortality. The incidence could be from 3.8 to5.5 episodes per 1000 days

Migration of micro-organism along the external surface of the catheter is probably the most common route of infection through skin and represents 58% .HD catheter has biofilm formation on their surfaces and this serves as a good reservoir for micro-organisms

Most patients with end stage renal disease (ESRD) starting hemodialysis through hemodialysis catheter about 9 % in Egypt and most of them require several hemodialysis catheters before maturation of arterio -venous fistula and even after stopping it.

DETAILED DESCRIPTION:
Patients receiving hemodialysis have a high risk of infection due to the immunosuppressive effects caused by ESRD, comorbidities, inadequate nutrition and the need for maintenance of vascular access for long periods.

The catheters are rightfully the least preferred modality and, in an ideal setting, no patient should have a catheter as access. Despite the perils associated with dialysis catheters, their use has increased to almost 70% incident dialysis initiation with catheters In dialysis centers, many patients are undergoing hemodialysis simultaneously, which facilitates the spread of microorganisms by direct or indirect contact through the devices, equipment, surface contact, and hands of health profession Over time, catheters are prone to higher rates of infection, thrombosis, and central venous stenosis, it has also been shown that catheters are an independent (of infection) inflammatory stressor and lead to increased morbidity Catheters are aptly referred to as a bacterial highway, and a biofilm formation around the catheter is often the breeding ground of bacteria and fungi, which can easily spread to the bloodstream Infectious complications are the most serious with regards to patient morbidity and mortality. The incidence could be from 3.8 to5.5 episodes per 1000 days

Migration of micro-organism along the external surface of the catheter is probably the most common route of infection through skin and represents 58% .HD catheter has biofilm formation on their surfaces and this serves as a good reservoir for micro-organisms

Most patients with end stage renal disease (ESRD) starting hemodialysis through hemodialysis catheter about 9 % in Egypt and most of them require several hemodialysis catheters before maturation of arterio -venous fistula and even after stopping it.

ELIGIBILITY:
Inclusion Criteria:

-Adults patients receiving long-term hemodialysis using temporary right internal jugular hemodialysis catheter

Exclusion Criteria:

* Age below 16
* Noncompliance patients
* Mechanical complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Catheter related infection | 45 days
  Catheter related infection which will manifest by fever rigor and obligatory remove of the catheter.

SECONDARY OUTCOMES:
The average duration of HD catheter | 45 days
  The average duration of HD catheter

CONTACTS AND LOCATIONS:
Overall Officials: Doaa ElBohy, PhD, Study Chair — FUE
Locations (1):
- Transplantation Clinic Nasser Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No